CLINICAL TRIAL: NCT06841848
Title: Fundus Camera Module for Early Detection of Alzheimer's Disease
Status: Recruiting | Type: Observational
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Responsible Party: Sponsor
Other Study IDs: CE/2023_023
Record Dates: First submitted 2025-02-17; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Ophthalmoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | US Export: No

GROUPS / COHORTS (2):
- Patients
  Interventions: Diagnostic Test: Fundoscopic Exam
- Healthy Subjects
  Interventions: Diagnostic Test: Fundoscopic Exam

INTERVENTIONS:
Diagnostic Test: Fundoscopic Exam — visualization of the retina using an ophthalmoscope

SUMMARY:
Alzheimer's Disease (AD) affects tens of millions of people just in Europe. It is typically detected in its late stage when irreversible damage has already occurred, and current treatments are mostly conservative or palliative. Here we developed a device performing high-resolution multispectral imaging of the eye fundus to detect AD in its early stage. After clinical testing, the proposed device has a high potential to become a method for routine population screening, as it is non-invasive and affordable. The possibility of AD detection in an early stage is crucial for developing a new pharmaceutical treatment that would dramatically improve the lives of millions and save the expenses connected to lifelong healthcare assistance to people with AD in later stages.

ELIGIBILITY:
Inclusion Criteria:

* 55 years or older
* Diagnosis:

  1. For AD group: Clinically diagnosed with Alzheimer's disease (mild to moderate stage) based on Mini-Mental State Examination (MMSE) score between 10-26 and confirmed by PET imaging or CSF.
  2. For Control group: No diagnosis of Alzheimer's disease or other neurodegenerative disorders.
* Signed informed consent by the patient. If there are any doubts that the patient is mentally capable of giving informed consent, the patient will be examined and verified to be mentally capable by an independent physician/ neurologist, prior to the initiation of any study specific procedure

Exclusion Criteria:

* Severe cognitive impairment (MMSE <10) preventing cooperation during the imaging process.
* Inability to remain still during the fundus imaging procedure.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is enrolled by Santa Lucia Foundation
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Validation of Multispectral Fundus Imaging for Alzheimer's Disease Detection | Baseline
  Create an automatic AD detection model using advanced data processing, such as machine learning, that would be able to distinguish between AD and a healthy retina.

CONTACTS AND LOCATIONS:
Locations (1):
- Santa Lucia Foundation, Rome, Italy, Italy